CLINICAL TRIAL: NCT05369728
Title: Medico-economic Evaluation of a Strategy With Coronary CT as First Line (CCTA) Compared With the Strategy With Functional Test as First Line, in Patients at Intermediate Risk of Developing Stable Coronary Disease.
Brief Title: Screening Of CoRonary ArTEry diSease
Acronym: SOCRATES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A00302-41
Record Dates: First submitted 2022-04-28; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Cardiology; Coronary Artery Disease
Keywords: Medico-economic study; Coronary CT scanner; Cardiac functionel test
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First line coronary scanner group (Other): The patient will benefit from a coronary CT scan in 1st line (evaluation of the coronary anatomy), then according to the result it will be managed according to the CAD-RADS decision algorithm.
  Interventions: Other: Coronary CT in 1st line compared to the strategy with functional test in 1st line in patient at Intermediate Risk of Developing Stable Coronary Disease:
- First line functional test strategy group (Other): The patient benefits from a functional test in 1st line (search for myocardial ischemia by myocardial scintigraphy: SPECT, stress echography, or MRI), then according to the result he will be managed in accordance with the European recommendations.
  Interventions: Other: Coronary CT in 1st line compared to the strategy with functional test in 1st line in patient at Intermediate Risk of Developing Stable Coronary Disease:

INTERVENTIONS:
Other: Coronary CT in 1st line compared to the strategy with functional test in 1st line in patient at Intermediate Risk of Developing Stable Coronary Disease: — Coronary CT in 1st line compared to the strategy with functional test in 1st line in Patients at Intermediate Risk of Developing Stable Coronary Disease:

SUMMARY:
This study is a randomized trial with the objective of comparing the cost-effectiveness of the 2 recommended strategies: CCTA vs functional tests, allowing the evaluation of the quality of life of these patients in relation to the health resources used.

In symptomatic patients with an intermediate probability of having stable CAD, i.e., whose pretest or clinical probability does not allow the elimination of the disease, and in patients without anginal symptoms for low levels of exercise who do not respond to medical therapy, in France, the diagnostic care pathways have become mature enough to set up a pragmatic prospective randomized trial with the objective of comparing the cost-effectiveness of the 2 recommended strategies: CCTA vs.

Probabilistic medico-economic reasoning makes it possible to establish this two-way hypothesis more easily than in clinical research without the need to impose the superiority of one of the strategies.

DETAILED DESCRIPTION:
In Europe, cardiovascular disease remains the leading cause of death with 4 million deaths per year, of which 1.8 million are due to coronary heart disease (CHD). CAD also has a cost with 46 billion / year spent for its management. In France, 4 billion are spent on it, which shows that it remains a public health problem and that most of the premature events are avoidable, in particular by screening patients with symptoms that make them suspect it. In these symptomatic patients suspected of having CAD, screening is carried out in particular through the use of imaging with technological innovations and performances that are constantly being improved and validated in large randomized trials.

The PROMISE trial randomized an impressive number of 10003 patients comparing coronary computed tomography angiography (CCTA) and functional testing to assess suspected CAD, which showed similar efficacy of the 2 strategies in terms of major adverse cardiovascular events (MACE) at 2 years: 3.3% for CCTA and 3% for functional testing. Thus, the 2019 European guidelines allow CCTA or functional testing as the initial test to diagnose CAD in symptomatic patients. Thus, clinicians now have 2 first-line strategies: CCTA or functional tests (myocardial scintigraphy, echocardiography, MRI). The clinician can choose to initiate management with an anatomic evaluation of the coronary arteries (CCTA) or a search for ischemia (functional test). These two ways of assessing CAD are very different and are the subject of debate in Europe. For example, the National Institute of Health and Care Excellence (NICE) in the United Kingdom now recommends CCTA as the first test, unlike in Europe.

In view of all these arguments, it is relevant to propose a randomized trial with the objective of comparing the cost-effectiveness of the 2 recommended strategies: CCTA vs. functional tests, making it possible to evaluate the quality of life of these patients in relation to the health resources used.

In symptomatic patients with an intermediate probability of having stable CAD, i.e., whose pretest or clinical probability does not allow the elimination of the disease, and in patients without anginal symptoms for low levels of exercise who do not respond to medical therapy, in France, the diagnostic care pathways have become mature enough to set up a pragmatic prospective randomized trial with the objective of comparing the cost-effectiveness of the 2 recommended strategies: CCTA vs.

Probabilistic medico-economic reasoning makes it possible to establish this two-way hypothesis more easily than in clinical research without the need to impose the superiority of one of the strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years
* Symptomatic patient in whom CAD cannot be excluded by clinical evaluation alone : patient with a pre-test or "intermediate" clinical probability indicating imaging test according to European recommendations
* Patient affiliated to the social security system or beneficiary of such a system
* Written informed consent

Exclusion Criteria:

* Pre-test probability "low" < 5% or 5-15% without additive pejorative factors
* Clinical probability of "high" CAD, defined by symptoms typical of low exercise levels not responding to medical therapies
* Known history of CAD
* Severe impairment of left ventricular ejection fraction < 40%.
* Known chronic renal failure not on dialysis (GFR <30 ml / min /1.73 m²)
* Patient considered unfit for the study according to the investigator's judgement and in particular the impossibility of performing an anatomical and/or functional test of ischemia of the coronary disease
* Patient in a period of exclusion for another study
* Persons referred to in articles L1121-5 to L1121-8 of the public health code
* Patient participating in another interventional research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Conduct a cost-utility analysis (CUA) comparing the strategy "CCTA in 1st line" to the strategy "functional test in 1st line" in patients with suspected stable CAD in a collective perspective, at 1 year. | 1 year
  The incremental cost-utility ratio (ICER) will be calculated by relating the difference in costs to the difference in the average number of QALYs. The ratio will therefore be expressed as cost per QALY gained, which represents the additional cost of gaining one year of healthy life with the "CCTA" strategy vs. the "functional test" strategy. Since CCTA is a special case of CEA, the incremental cost-effectiveness ratio (ICER) expressed as the incremental cost per life-year gained will also be calculated.

SECONDARY OUTCOMES:
To model in the long term (10 years) the impact of the 2 diagnostic strategies in terms of cost and consequences as defined in the main objective. | 10 years
  Incremental cost-effectiveness ratio (ICER and ICER) at 10 years as defined in Primary Objective 1.
Conduct a budget impact analysis (BIA) from the National Health System's perspective at 3 and 5 years. | 3 and 5 years
  Measure the financial impact on the National Health System of the deployment of the CCTA strategy in 3 and 5 years
To compare angina symptoms (limitation, stability, frequency) at 1 year. | 1 year
  SAQ (Seattle Angina Questionnaire): physical limitation is assessed by question 1; angina stability by question 2 and angina frequency by questions 3 and 4
Compare treatment satisfaction at 1 year | 1 year
  SAQ: patients' satisfaction with their current treatment is assessed in questions 5 to 8
Compare quality of life at 1 year | 1 year
  SAQ: quality of life is assessed in questions 9 to 11 of the questionnaire
Compare dyspnea at 1 year | 1 year
  ROSE dyspnea scale : grade 1 to 4 (worst condition)
Compare severity of angina at 1, 2 and 3 years | 1, 2 and 3 years
  CCS score (Canadian Cardiovascular Society) : grade asymptomatic to 4 (worst condition)
Compare quality of life at 1, 2 and 3 years | 1, 2 and 3 years
  Quality of life: EuroQol 5D-5 : cotation from 0 (worst condition) to 1.
Compare the care pathways of the "CCTA" strategy to the "Functional Test" strategy at 1 year. | 1 year
  Number of CAD imaging tests
Compare the care pathways of the "CCTA" strategy to the "Functional Test" strategy at 1 year. | 1 year
  Time to obtain CAD imaging tests
Compare the care pathways of the "CCTA" strategy to the "Functional Test" strategy at 1 year. | 1 year
  Type of CAD imaging tests
Compare the care pathways of the "CCTA" strategy to the "Functional Test" strategy at 1 year. | 1 year
  Treatments used after the first line examination to manage chest pain symptomatology
Observe deviations in management from current recommendations at 1 year. | 1 year
  Number and percentage of deviations from current recommendations
Compare the diagnostic benefit of the CCTA strategy to the Functional Test strategy at 1 year. | 1 year
  Number and rate of coronary angiography with or without FFR/iwFR
Compare the diagnostic benefit of the CCTA strategy to the Functional Test strategy at 1 year. | 1 year
  Number and rate of revascularization
Compare major clinical events at 1, 2 and 3 years. | 1, 2 and 3 years.
  Deaths from cardiovascular causes, myocardial infarction, or ischemia-guided revascularization, heart failure, or recovered cardiac arrest.
Compare the radiation exposure of patients for each strategy at 1 year. | 1 year
  Measurement of radiation exposure related to cardiovascular tests and procedures in millisieverts
To study the influence of new indexes from post image processing on the consumption of care and on the symptoms of angina. | 1 year
  New indexes from post image processing
To study the influence of new indexes from post image processing on the consumption of care and on the symptoms of angina. | 1 year
  QUALY
To study the influence of new indexes from post image processing on the consumption of care and on the symptoms of angina. | 1 year
  SAQ (Seattle Angina questionnaire) question 1 to 19

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Barone-Rochette, Pr, Principal Investigator — CHU Grenoble Alpes

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Roth GA, Johnson C, Abajobir A, Abd-Allah F, Abera SF, Abyu G, Ahmed M, Aksut B, Alam T, Alam K, Alla F, Alvis-Guzman N, Amrock S, Ansari H, Arnlov J, Asayesh H, Atey TM, Avila-Burgos L, Awasthi A, Banerjee A, Barac A, Barnighausen T, Barregard L, Bedi N, Belay Ketema E, Bennett D, Berhe G, Bhutta Z, Bitew S, Carapetis J, Carrero JJ, Malta DC, Castaneda-Orjuela CA, Castillo-Rivas J, Catala-Lopez F, Choi JY, Christensen H, Cirillo M, Cooper L Jr, Criqui M, Cundiff D, Damasceno A, Dandona L, Dandona R, Davletov K, Dharmaratne S, Dorairaj P, Dubey M, Ehrenkranz R, El Sayed Zaki M, Faraon EJA, Esteghamati A, Farid T, Farvid M, Feigin V, Ding EL, Fowkes G, Gebrehiwot T, Gillum R, Gold A, Gona P, Gupta R, Habtewold TD, Hafezi-Nejad N, Hailu T, Hailu GB, Hankey G, Hassen HY, Abate KH, Havmoeller R, Hay SI, Horino M, Hotez PJ, Jacobsen K, James S, Javanbakht M, Jeemon P, John D, Jonas J, Kalkonde Y, Karimkhani C, Kasaeian A, Khader Y, Khan A, Khang YH, Khera S, Khoja AT, Khubchandani J, Kim D, Kolte D, Kosen S, Krohn KJ, Kumar GA, Kwan GF, Lal DK, Larsson A, Linn S, Lopez A, Lotufo PA, El Razek HMA, Malekzadeh R, Mazidi M, Meier T, Meles KG, Mensah G, Meretoja A, Mezgebe H, Miller T, Mirrakhimov E, Mohammed S, Moran AE, Musa KI, Narula J, Neal B, Ngalesoni F, Nguyen G, Obermeyer CM, Owolabi M, Patton G, Pedro J, Qato D, Qorbani M, Rahimi K, Rai RK, Rawaf S, Ribeiro A, Safiri S, Salomon JA, Santos I, Santric Milicevic M, Sartorius B, Schutte A, Sepanlou S, Shaikh MA, Shin MJ, Shishehbor M, Shore H, Silva DAS, Sobngwi E, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadele Atnafu N, Tesfay F, Thakur JS, Thrift A, Topor-Madry R, Truelsen T, Tyrovolas S, Ukwaja KN, Uthman O, Vasankari T, Vlassov V, Vollset SE, Wakayo T, Watkins D, Weintraub R, Werdecker A, Westerman R, Wiysonge CS, Wolfe C, Workicho A, Xu G, Yano Y, Yip P, Yonemoto N, Younis M, Yu C, Vos T, Naghavi M, Murray C. Global, Regional, and National Burden of Cardiovascular Diseases for 10 Causes, 1990 to 2015. J Am Coll Cardiol. 2017 Jul 4;70(1):1-25. doi: 10.1016/j.jacc.2017.04.052. Epub 2017 May 17. PMID 28527533
- [Background] Timmis A, Townsend N, Gale CP, Torbica A, Lettino M, Petersen SE, Mossialos EA, Maggioni AP, Kazakiewicz D, May HT, De Smedt D, Flather M, Zuhlke L, Beltrame JF, Huculeci R, Tavazzi L, Hindricks G, Bax J, Casadei B, Achenbach S, Wright L, Vardas P; European Society of Cardiology. European Society of Cardiology: Cardiovascular Disease Statistics 2019. Eur Heart J. 2020 Jan 1;41(1):12-85. doi: 10.1093/eurheartj/ehz859. PMID 31820000
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439